CLINICAL TRIAL: NCT00188331
Title: Cognitive Function and Fatigue in Cancer Patients After Chemotherapy: A Longitudinal Controlled Study in Patients With Colorectal Cancer
Brief Title: Cognitive Function and Fatigue in Colorectal Cancer (CRC) Patients After Chemotherapy
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Cancer Trials Group (Network); Young Investigator Award - American Society of Clinical Oncologists (Unknown); Peterborough K.M. Hunter Graduate Studentship (Unknown)
Responsible Party: Sponsor
Other Study IDs: COIT1; NCIC Grant No. #15261
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Cognition; Fatigue; Colorectal Neoplasm
Keywords: cognitive function; fatigue; colorectal cancer; chemotherapy; cognitive impairment
MeSH Terms: conditions — Fatigue; Colorectal Neoplasms; Cognitive Dysfunction | interventions — Neuropsychological Tests

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — cytokines, genotyping apoE, EUC, LFTs, sex hormones, coagulation factors
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: adjuvant/neoadjuvant chemotherapy
  Interventions: Behavioral: Neuropsychological Testing
- 2: non-chemotherapy group
  Interventions: Behavioral: Neuropsychological Testing
- 3: limited metastatic disease or localised recurrence to receive first line metastatic chemotherapy
  Interventions: Behavioral: Neuropsychological Testing

INTERVENTIONS:
Behavioral: Neuropsychological Testing — neuropsychological testing with traditional tests, CANTAB and six elements test as well as questionnaires

SUMMARY:
This is a prospective, longitudinal cohort study to evaluate fatigue and cognitive function in patients with colorectal cancer (CRC) treated with chemotherapy, and in patients with the same malignancy, that do not receive chemotherapy. A self-report questionnaire for fatigue (the FACT-F), and validated tests of cognitive function, will be applied at predetermined times before, during and after chemotherapy, to determine the incidence, severity and duration of these symptoms. Comparisons will be made in changes in cognition for individuals, as well as between the chemotherapy and the control group. Mechanisms that might lead to fatigue and/or cognitive decline will be investigated.

DETAILED DESCRIPTION:
We will undertake a prospective, longitudinal controlled study of fatigue and cognitive function in 120 patients with localized CRC who receive 5FU-based adjuvant chemotherapy. Each patient will be evaluated at baseline and at 6, 12 and 24 months for fatigue (using the FACT-F questionnaire) and for cognitive function, using validated tests: these will comprise both traditional neuropsychological tests and the computerised CANTAB™, a which is less dependent on fluency in English. Results during and after chemotherapy will be compared with the pre-chemotherapy assessment (so that each patient acts as their own control). Since baseline evaluation may be confounded by the recent diagnosis and surgery we will include an independent control group of 120 patients who have undergone surgery for CRC but who do not receive chemotherapy. Patients found to have cognitive change will be offered further comprehensive neuropsychological assessment. We will also evaluate quality of life (QOL) using the FACT-G questionnaire and anxiety and depression using the General Health Questionnaire (GHQ). Blood tests including hormone levels, cytokines, homocysteine, procoagulants and apo-lipoprotein E-є4 allele status will evaluate possible mechanisms. Finally, since chemotherapy for CRC is evolving to include the more toxic drugs oxaliplatin and irinotecan, we will perform a parallel pilot study evaluating pts with early recurrent or metastatic CRC who receive these drugs, using similar methods of evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed colorectal cancer
* Age 18-75
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Life expectancy of at least 12 months
* Full recovery from any post operative sequelae
* Adequate hepatic function as documented by a serum bilirubin < 18 umol/L, and liver function tests (LFTs) within 1.5X normal range
* Informed consent

Exclusion Criteria:

* Any major pre-existing psychiatric history or dementia, alcohol abuse, or currently using a psychotropic medication that might lead to cognitive problems, other than short acting benzodiazepines for nausea or sleep
* Any evidence of metastatic disease other than group C who may have limited metastatic disease. If there is clinical suspicion of central nervous system (CNS) involvement patients must have brain imaging (MRI or CT scan) prior to recruitment.
* Ongoing sepsis or uncontrolled infection, including HIV infection
* Pre-existing neurological condition likely to interfere with ability to perform cognitive testing
* Any other severe co-morbidity which, in the judgement of the investigator, would make the patient inappropriate for entry into this study
* Active cancer within the last 5 years other than squamous or basal cell carcinoma of the skin or cervical cancer in situ (except for CRC)
* Previous history of chemotherapy, other than adjuvant chemotherapy for group C metastatic group > 1 year previously
* Minimal English skills such that subjects would be unable to follow simple, written English instructions and to read questionnaires of a grade 8 standard with the help of a research assistant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: colorectal cancer patients aged 18-75
Sampling Method: Probability Sample
Enrollment: 441 (Actual)
Dates: Start 2003-11; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janette Vardy, MD, Principal Investigator — Princess Margaret Hospital University of Toronto; Ian Tannock, Principal Investigator — Princess Margaret Hospital University of Toronto
Locations (2):
- Sydney Cancer Centre, Sydney, New South Wales, Australia
- University Health Network, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Vardy JL, Dhillon HM, Pond GR, Renton C, Clarke SJ, Tannock IF. Prognostic indices of inflammatory markers, cognitive function and fatigue for survival in patients with localised colorectal cancer. ESMO Open. 2018 Feb 14;3(2):e000302. doi: 10.1136/esmoopen-2017-000302. eCollection 2018. PMID 29531839
- [Derived] Dhillon HM, Tannock IF, Pond GR, Renton C, Rourke SB, Vardy JL. Perceived cognitive impairment in people with colorectal cancer who do and do not receive chemotherapy. J Cancer Surviv. 2018 Apr;12(2):178-185. doi: 10.1007/s11764-017-0656-6. Epub 2017 Oct 27. PMID 29080061
- [Derived] Vardy JL, Dhillon HM, Pond GR, Renton C, Dodd A, Zhang H, Clarke SJ, Tannock IF. Fatigue in people with localized colorectal cancer who do and do not receive chemotherapy: a longitudinal prospective study. Ann Oncol. 2016 Sep;27(9):1761-7. doi: 10.1093/annonc/mdw252. Epub 2016 Jul 20. PMID 27443634
- [Derived] Vardy J, Dhillon HM, Pond GR, Rourke SB, Xu W, Dodd A, Renton C, Park A, Bekele T, Ringash J, Zhang H, Burkes R, Clarke SJ, Tannock IF. Cognitive function and fatigue after diagnosis of colorectal cancer. Ann Oncol. 2014 Dec;25(12):2404-2412. doi: 10.1093/annonc/mdu448. Epub 2014 Sep 11. PMID 25214544